CLINICAL TRIAL: NCT05557188
Title: The Effect of Grounding on Leg Cramps, Sleep, Fatigue, Anxiety, and Quality of Life During Pregnancy
Brief Title: The Effect of Grounding During Pregnancy
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Ege University (Other)
Responsible Party: Principal Investigator, Esma Yuksel, Research assistant at the Faculty of Health Sciences, Ege University. Midwife, MSc., PhD. (Candidate), Ege University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 20-4T/39
Record Dates: First submitted 2022-09-19; First posted 2022-09-27 (Actual); Last update posted 2023-05-01 (Actual); Status verified 2023-04

CONDITIONS: Cramp, Limb; Pregnancy Related
Keywords: Cramp, Fatigue, Pregnancy
MeSH Terms: conditions — Muscle Cramp; Fatigue

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Sham Grounding (Placebo Comparator): Each pregnant woman in the placebo group is going to be informed about the Sham grounding stick and how to use it, with a 2-minute video showing. Participants walk on the ground for 30 minutes daily and go on for four weeks. During the program, the pregnant women will be called to their homes every week and necessary reminders will be made.
  Interventions: Other: Sham grounding
- Grounding (Active Comparator): Each pregnant woman in the placebo group is going to be informed about the grounding stick and how to use it, with a 2-minute video showing. Participants walk on the ground for 30 minutes daily and go on for four weeks. During the program, the pregnant women will be called to their homes every week and necessary reminders will be made.
  Interventions: Other: Grounding

INTERVENTIONS:
Other: Grounding — Each pregnant woman in the placebo group is going to be informed about the grounding stick and how to use it, with a 2-minute video showing. Participants walk on the ground for 30 minutes daily and go on for four weeks. During the program, the pregnant women will be called to their homes every week and necessary reminders will be made.
  Arms: Grounding
Other: Sham grounding — Each pregnant woman in the placebo group is going to be informed about the Sham grounding stick and how to use it, with a 2-minute video showing. Participants walk on the ground for 30 minutes daily and go on for four weeks. During the program, the pregnant women will be called to their homes every week and necessary reminders will be made.
  Arms: Sham Grounding

SUMMARY:
The study was planned as a randomized controlled trial. The research data included a pregnant informed form, leg cramps evaluation form, Pittsburgh Sleep Quality Index, Visual Analog Scale for fatigue, Pregnancy-Related Anxiety Scale, Short Form-12 Quality of Life Scale, food consumption record form, and pregnancy follow-up form will be used. Questionnaires will be evaluated every two weeks, and the intervention will continue for four weeks in total for each pregnant woman.

DETAILED DESCRIPTION:
The aim of the research is to investigate the effect of grounding on muscle cramps, sleep quality, fatigue, anxiety, and quality of life in pregnant women. The study was planned as a randomized controlled trial. The study is going to perform in the Obstetrics and Gynecology Clinic of Ege University Medical Faculty Hospital. The research will be carried out by face-to-face interview method. The research data included a pregnant informed form, leg cramps evaluation form, Pittsburgh Sleep Quality Index, Visual Analog Scale for fatigue, Pregnancy-Related Anxiety Scale, Short Form-12 Quality of Life Scale, food consumption record form, and pregnancy follow-up form will be used. The pregnant women included in the study will be divided into two groups as intervention and placebo groups by randomization and will be asked to take a walk for 30 minutes every day with a grounding/sham grounding pole. Questionnaires will be evaluated every two weeks, and the intervention will continue for four weeks in total for each pregnant woman.

ELIGIBILITY:
Inclusion Criteria:

* Between 27-34 weeks of pregnancy,
* Having leg cramps,
* Normal blood levels of calcium and magnesium in her current pregnancy,
* No risky pregnancy, or chronic disease (heart disease, hypertension, thyroid diseases, diabetes mellitus, kidney disease, etc.)
* Not having multiple pregnancies,

Exclusion Criteria:

* Risky pregnancy, chronic disease (heart disease, hypertension, thyroid diseases, diabetes mellitus, kidney disease, etc.),
* Emerging Rheumatic Disease,
* Varicose veins in the legs,
* Diagnosed with restless legs syndrome,
* Pregnant women with blood levels of Calcium and Magnesium below the normal level will be excluded from the study.

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — In this study, pregnant women are going to enroll.
Enrollment: 86 (Estimated)
Dates: Start 2022-11-01 (Actual); Primary Completion 2023-11-01 (Estimated); Study Completion 2024-02-01 (Estimated)

PRIMARY OUTCOMES:
Pittsburgh Sleep Quality Index | 10 minutes.
  It is a safe and consistent sleep questionnaire that includes 24 questions to evaluate sleep quality, amount of sleep, presence and severity of sleep disorder in the last month.
Leg Cramps Evaluation Form | 3 minutes.
  There are questions about the duration and frequency of leg cramps, what has been done to relieve the pain and the Visual Analog Scale that will be used to assess the pain in leg cramps. Higher scores mean worse outcome.

SECONDARY OUTCOMES:
Visual analog scale for Fatigue | 12 minutes
  The scale consists of two categories: fatigue (items 1, 2, 3, 4, 5, 11, 12, 13, 14, 15, 16, 17, 18) and energy (items 6, 7, 8, 9, 10). It consists of sub-dimensions and 18 items. There are 10 cm long horizontal lines with positive words on one end of the scale and negative words on the other.
Pregnancy-Related Anxiety Scale | 8 minutes.
  The 11-item questionnaire was structured in three dimensions: fear of giving birth (items 1, 2, 6 and 8), concerns about carrying a disabled child (items 4, 9, 10 and 11) and concerns about your own appearance (3, 5 and 7). ) contains. The eighth item of the questionnaire ("I am worried about childbirth because I have never experienced it before") applies only to primiparous women. Items are rated from 1-5 (1 = "not at all relevant" and 5 = "very relevant"). Higher scores mean a worse outcome.
Short Form-12 Quality of Life Scale | 12 minutes.
  It consists of 12 questions selected from the SF-36 Health Questionnaire. SF-12 consists of physical functionality, physical role, pain, general health, emotional role, social functionality and vitality subcomponents.

CONTACTS AND LOCATIONS:
Overall Officials: Esma YUKSEL, Principal Investigator — Ege University
Locations (2):
- Turkey (Türkiye) (2):
  - Ege University, Izmir
  - Murat Pehlivan, Izmir

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Allen RE, Kirby KA. Nocturnal leg cramps. Am Fam Physician. 2012 Aug 15;86(4):350-5. PMID 22963024
- [Result] Chevalier G, Sinatra ST, Oschman JL, Delany RM. Earthing (grounding) the human body reduces blood viscosity-a major factor in cardiovascular disease. J Altern Complement Med. 2013 Feb;19(2):102-10. doi: 10.1089/acm.2011.0820. Epub 2012 Jul 3. PMID 22757749
- [Result] Brown D, Chevalier G, Hill M. Pilot study on the effect of grounding on delayed-onset muscle soreness. J Altern Complement Med. 2010 Mar;16(3):265-73. doi: 10.1089/acm.2009.0399. PMID 20192911